CLINICAL TRIAL: NCT06710860
Title: An Intelligent Voice-interactive Tailored Communication System (ScreenTalk) for Enhancing Colorectal Cancer Screening Among First-degree Relatives of Patients: a Randomized Type I Hybrid Effectiveness-implementation Trial
Brief Title: ScreenTalk to Improve Colorectal Cancer Screening Uptake Among First-degree Relatives of Patients: a Study Protocol
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: National Natural Science Foundation of China (Other Government)
Responsible Party: Principal Investigator, Yang Bai, Associate Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: L2024SYSU-HL-054
Record Dates: First submitted 2024-11-26; First posted 2024-11-29 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-11

CONDITIONS: Colonoscopy; Colorectal Cancer; First-degree Relatives
Keywords: Colonoscopy; First-degree relatives; Cancer screening; Artificial intelligence; Speech technology; Type I hybrid effectiveness-implementation trial; RE-AIM framework
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): ScreenTalk AI-based tailored communication intervention
  Interventions: Behavioral: The intelligent voice-interactive tailored communication system-based intervention
- Attention control group (No Intervention): Targeted communication, attention control

INTERVENTIONS:
Behavioral: The intelligent voice-interactive tailored communication system-based intervention — Participants in intervention group will receive the ScreenTalk intervention consisting of 3 modules:(1) a measurement module, (2) an algorithmic tailoring module, and (3) an open di-alogue module. All participants will be required to complete 3 modules within 1 month. If the intervention group does not undergo CRC screening at the follow-up time point, the system will repeatedly provide tailored communication intervention to further enhance the CRC risk perception of FDRs based on the current evaluation results. The primary outcome (uptake of CRC screening) will be measured at 3 months post-intervention (T1), 6 months post-intervention (T2), 9 months post-intervention (T3) and 12 months post-intervention (T4).
  Arms: Intervention group

SUMMARY:
Participants in intervention group will receive the ScreenTalk intervention consisting of 3 module: measurement module, algorithmic tailoring module, and open dialogue module. The primary outcome, CRC screening uptake will be verified by medical records; and health belief will be measured at baseline, 3, 6, 9 and 12 months.

DETAILED DESCRIPTION:
This study will follow a hybrid type I effectiveness-implementation trial design. A cluster-randomized controlled trial will be conducted to examine the effectiveness of the intelligent voice-interactive tailored communication system. ScreenTalk can automatically tailor screening recommendations based on risk and psychosocial characteristic assessments by leveraging intelligent speech interaction (ISI) technology. The three components of the ScreenTalk intervention are as follows: (1) a measurement module, (2) an algorithmic tailoring module, and (3) an open dialogue module. All participants will be required to complete 3 modules within 1 month. If the intervention group does not undergo CRC screening at the follow-up time point, the system will repeatedly provide tailored communication intervention to further enhance the CRC risk perception of FDRs based on the current evaluation results. The implementation outcomes will be guided by the RE-AIM framework. Both qualitative and quantitative methods will be employed to evaluate implementation outcomes and determine the factors that may influence implementation process. CRC screening uptake verified by medical records and health belief will be measured at baseline, 3, 6, 9 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 75 years or 10 years before the age at which the relative was diagnosed;
* individuals with one FDR with CRC age <60 years or with two or more FDRs with CRC at any age;
* have not had a colonoscopy within 5 years;
* access to WeChat themselves or through close family members living in the same household;
* able to read and speak Chinese.

Exclusion Criteria:

* Have history of cancer or inflammatory bowel disease;
* have history of a hereditary syndromes (Lynch syndrome or familial adenomatous polyposis);
* recently participate in another study or previously participated in cancer risk counseling or study;
* with doctor-diagnosed psychiatric illness.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Participate rate of CRC screening | 3 months post-intervention (T1); 6 months post-intervention (T2); 9 months post-intervention (T3); 12 months post-intervention (T4)
  Uptake of colonoscopy or FOBT. Medical records will be collected from those who had undergone colonoscopy or fecal test. Only the examination records that are verified by medical records will be counted and involved in the data analysis.

SECONDARY OUTCOMES:
Perceived threat | Baseline (T0); 3 months post-intervention (T1); 6 months post-intervention (T2); 9 months post-intervention (T3); 12 months post-intervention (T4)
  The Colorectal Cancer and Colonoscopy Screening Health Beliefs Scale for First-Degree Relatives (CCHBS-FDR), with 6 dimensions, will be used to measures perceived threat of CRC and colonoscopy screening, namely per-ceived susceptibility of CRC and perceived severity of CRC. Each item of CCHBS-FDR is rated on a five-point (1-5) Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree), with scores ranging from 36 to 180. Higher scores on each dimension indicate higher levels of perception.
Perceived efficacy | Baseline (T0); 3 months post-intervention (T1); 6 months post-intervention (T2); 9 months post-intervention (T3); 12 months post-intervention (T4)
  Perceived efficacy includes perceived benefits and self-efficacy. The Colorectal Cancer and Colonoscopy Screening Health Beliefs Scale for First-Degree Relatives (CCHBS-FDR) will be used to measures perceived efficacy of colonoscopy screening, and the four-item simplified Chinese version of the self-efficacy questionnaire will be used to assess the self-efficacy for participating in CRC screening. Each item of these two questionnaires is rated on a five-point (1-5) Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree), with scores ranging from 36 to 180. Higher scores on each dimension indicate higher levels of perception.
Perceived barriers | Baseline (T0); 3 months post-intervention (T1); 6 months post-intervention (T2); 9 months post-intervention (T3); 12 months post-intervention (T4)
  The Colorectal Cancer and Colonoscopy Screening Health Beliefs Scale for First-Degree Relatives (CCHBS-FDR) will be used to measures perceived barriers for participating in CRC screening. Each item of CCHBS-FDR is rated on a five-point (1-5) Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree), with scores ranging from 36 to 180. Higher scores on each dimension indicate higher levels of perception.
Cue to action | Baseline (T0); 3 months post-intervention (T1); 6 months post-intervention (T2); 9 months post-intervention (T3); 12 months post-intervention (T4)
  Including three types of action cues: family history of CRC, physician's recommendation and health insurance coverage. The cue to action for CRC screening questionnaire will be used to collect information of cue to action among FDRs. Each item is rated on a five-point (1-5) Likert scale ranging from 1 (Strongly Disagree) to 5 (Strongly Agree). The score for cues to action was calculated by averaging the corresponding items (ranging from 1 to 5), with higher score indi-cating higher cue to action.

OTHER OUTCOMES:
Participant characteristics | Baseline (T0)
  A self-designed general information questionnaire will be used to collect participant characteristics.
Percentage of contacted FDRs who participate in this study | Baseline (T0); 1 month post-intervention
  Collect data through information recorded in the Implementation logbook
Enrollment routes | Baseline (T0)
  Including the recruitment approach and reasons for refusal to participate. It will be collected through the implementation logbook.
Representativeness of staff that participate | Baseline (T0)
  The self-designed general information questionnaire for staff will be used to collect related data.
Barriers and facilitators to adoption | 13 months post-intervention
  Qualitative interviews will be conducted to gain staff insights into intervention adoption.
Fidelity | 1 month post-intervention; post-implementation
  Fidelity includes participants' adherence of each module and reasons for non-completion. Relevant data will be collected through the tailored communication system record.
Acceptability | 1-month post intervention
  The User Feedback Questionnaire for ScreenTalk will be used to measure the satisfaction among the participant for ScreenTalk.
Maintenance | 3 months post-intervention (T1); 6 months post-intervention (T2); 9 months post-intervention (T3); 12 months post-intervention (T4)
  Sustained engagement of participants at 3-month, 6-month, 9-month, and 12-month follow-up. Follow-up information of participants will be obtained through the implementation logbook and tailored communication system record.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - The Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lin S, Luo B, Cai L, Qiu L, Li H, Liu W, Luo Y, Yuan Y, Peng Z, Bai Y. Intelligent voice-interactive tailored communication system (ScreenTalk) to improve colorectal cancer screening uptake among first-degree relatives of colorectal cancer patients: study protocol for a cluster-randomised type I hybrid effectiveness-implementation trial. BMJ Open. 2025 Dec 10;15(12):e109534. doi: 10.1136/bmjopen-2025-109534. PMID 41371735